CLINICAL TRIAL: NCT04972942
Title: Phase I Trial of Targeted Immunotherapy with Daratumumab Following Myeloablative TBI-Based Conditioning and AlloHCT in Children, Adolescents and Young Adults with High Risk T-Cell Acute Lymphoblastic Leukemia and Lymphoma (ALLO-T-DART)
Brief Title: Targeted Immunotherapy After Myeloablative TBI-Based Conditioning & AlloHCT in CAYA with High Risk T-Cell ALL & Lymphoma
Acronym: ALLO-T-DART
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-598
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; T-Cell Acute Lymphoblastic Lymphoma
Keywords: immunotherapy; children; adolescents; young adults
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Phase 1: 3 dose levels to determine safety. Followed by dose expansion cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional (Other): Phase 1: 3 dose levels to determine safety (15 patients)
  Dose expansion:
  Daratumumab (DARA) treatment post-HCT
  1. Induction: DARA IV weekly x 8 doses (Weeks 1-8)
  2. Consolidation: DARA IV every 2 weeks x 8 doses (Weeks 9-24)
  3. Maintenance: DARA IV every 4 weeks (Stop at Day +270)
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Total body irradiation (TBI)-based myeloablative allogeneic hematopoietic stem cell transplantation (HCT) using best available donor.
  Daratumumab (DARA) treatment post-HCT Phase 1: 3 dose levels to determine safety (15 patients)
  Dose expansion:
  1. Induction: DARA IV weekly x 8 doses (Weeks 1-8)
  2. Consolidation: DARA every 2 weeks x 8 doses (Weeks 9-24)
  3. Maintenance: DARA every 4 weeks (Stop at Day +270)
  Other Names: Darzalex®

SUMMARY:
A Phase I trial to determine the safety of targeted immunotherapy with daratumumab (DARA) IV after total body irradiation (TBI)-based myeloablative conditioning and allogeneic hematopoietic cell transplantation (HCT) for children, adolescents, and young adults (CAYA) with high risk T-cell acute lymphoblastic leukemia (T-ALL) or T-cell lymphoblastic lymphoma (T-LLy).

Pre- and post-HCT NGS-MRD studies will be correlated with outcomes in children, adolescents, and young adults with T-ALL undergoing allogeneic HCT and post-HCT DARA treatment. The study will also evaluate T-cell repertoire and immune reconstitution prior to and following DARA post-HCT treatment and correlate with patient outcomes.

DETAILED DESCRIPTION:
Total body irradiation (TBI)-based myeloablative allogeneic hematopoietic stem cell transplantation (HCT) using best available donor.

Daratumumab (DARA) treatment post-HCT:

Phase 1: 3 dose levels to determine safety (15 patients)

Dose expansion cohort (DEC): Further evaluation of PK and PD (correlative studies/exploratory endpoints) to guide future selection of RP2D (15 patients)

Treatment Schedule:

1. Induction: DARA IV weekly x 8 doses (Weeks 1-8)
2. Consolidation: DARA IV every 2 weeks x 8 doses (Weeks 9-24)
3. Maintenance: DARA IV every 4 weeks (Stop at Day +270)

ELIGIBILITY:
Inclusion Criteria:

* 0-39yrs
* T-cell ALL in second or subsequent remission (≤ 5% blasts) or relapsed T-cell LLy with complete response after re-induction therapy (including secondary malignancy)
* Planned allogeneic stem cell transplantation with donor identified
* Performance status ≥ 60%
* Fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Meet organ function requirements
* Signed IRB approved informed consent

Exclusion Criteria:

* May not have had a prior autologous or allogenic stem cell transplant
* May not have uncontrolled, systemic infection at the time of enrollment
* Known allergies, hypersensitivity, or intolerance to mannitol, sorbitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients
* Must not be pregnant or actively breast feeding
* Seropositive for HIV, hepatitis B or hepatitis C
* COPD
* Asthma
* Clinically significant cardiac disease

Max Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Patients with dose limiting toxicity (per CTCAE v.5) | 60 days
  occurrence of any Grade ≥ 3 non hematologic toxicity (per CTCAE v.5) which is probably, or definitely related to daratumumab

SECONDARY OUTCOMES:
Relapse free survival | 1 year
  To measure relapse free survival in patients post HCT and daratumumab

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Study Chair — New York Medical College; Troy Quigg, DO, Study Chair — Helen DeVos Children's Hospital; Allyson Flower, MD, Study Chair — New York Medical College
Locations (16):
- United States (16):
  - Phoenix Children's Hospital, Phoeniz, Arizona
  - Loma Linda University Children's Hospital, Loma Linda, California
  - University of California, Los Angeles, California
  - University of California, San Francisco, California
  - Children's Hospital Colordao, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainsville, Florida
  - John Hopkins All Children's Hospital, St. Petersburg, Florida
  - Riley Children's Hospital, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - New York Medical College, Vallhala, New York
  - Nationwide Children's Hosptial, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No